CLINICAL TRIAL: NCT03293862
Title: Prevention of Fascial Dehiscence With Prophylactic Onlay Mesh in Emergency Laparotomies: a Randomized Clinical Trial
Brief Title: Prevention of Fascial Dehiscence With Prophylactic Onlay Mesh in Emergency Laparotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Edivaldo Massazo Utiyama, MD, PhD, Full Professor of Surgery, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024878
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Surgical Wound Dehiscence
Keywords: laparotomy; emergency surgery; abdominal wound dehiscence; prophylactic mesh
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: Suture group and prophylactic mesh group
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suture group (Active Comparator): Patients randomized to this arm will undergo midline laparotomy closure using a PDS 0 continuous suture only, without mesh, aiming a suture length to wound length ratio higher than four. Randomization occurs after fascial closure.
  Interventions: Procedure: Midline Fascial Closure
- Prophylactic mesh group (Experimental): Patients randomized to this arm will undergo midline laparotomy closure using a PDS 0 continuous suture aiming a suture length to wound length ratio higher than four AND further polypropilene onlay mesh. Randomization occurs after fascial closure.
  Interventions: Device: prophylactic polypropilene mesh; Procedure: Midline Fascial Closure; Device: vacuum drainage system

INTERVENTIONS:
Device: prophylactic polypropilene mesh — Placement of onlay polypropilene prophylactic mesh after midline fascial closure.
  Arms: Prophylactic mesh group
Procedure: Midline Fascial Closure — midline fascial closure using uninterrupted PDS 0 suture
Device: vacuum drainage system — Placement of a subcutaneous vacuum drainage system
  Arms: Prophylactic mesh group

SUMMARY:
Facial dehiscence elicit high morbidity and mortality. This complication may arise in more than 8.5% of high-risk patients. Addressing risk factors and optimizing surgical technique are guarded as mainstay measures for prevention, but their efficacy is questionable. The aim of this study is to analyze the influence of using a polypropylene onlay prophylactic mesh on the incidence of fascial dehiscence in emergency surgery and associated complications.

DETAILED DESCRIPTION:
Fascial dehiscence is associated with high morbidity and mortality rates. It occurs in more than 8.5% of high-risk patients. Current preventive measures described are control of risk factors and optimization of surgical technique. Despite that, the incidence of such complication remained stable in the last decades, highlighting the low efficacy of such measures. Polypropilene onlay mesh has been used to avoid incisional hernias in selected elective patients, and could be useful in the prevention of fascial dehiscence. In emergency situations, especially in contaminated and infected surgical procedures, safety and efficacy of mesh is controversial. In this study the investigators aimed to evaluate the influence of polypropilene prophylactic onlay mesh on the incidence of fascial dehiscence in high-risk patients undergoing midline emergency laparotomy. As secondary outcome, the associated morbidity, including surgical site occurence, will be analyzed. The study design will be a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Emergency laparotomy by midline incision
* High risk for abdominal wound dehiscence: Risk index** ≥ 4,0 or ≥ 2,2 in combination with at least one of the following: smoking, obesity, malnutrition or malignant neoplasia.

  * Risk index is the sum of values associated with high-risk characteristics, based in the risk score for abdominal wall dehiscence published by van Ramshorst et. al. in World Journal of Surgery, 2010 (Rotterdam risk model):

Age category (in years)

* 40-49: 0.4
* 50-59: 0.9
* 60-69: 0.9
* ≥70: 1.1

Male gender: 0.7

Chronic pulmonary disease: 0.7

Ascites: 1.5

Jaundice: 0.5

Anemia: 0.7

Emergency surgery: 0.6

Type of surgery:

* Gallbladder/bile duct 0.7
* Esophagus 1.5
* Gastroduodenum 1.4
* Small bowel 0.9
* Large bowel 1.4
* Vascular 1.3

Exclusion Criteria:

* Non-midline incisions or midline laparotomy measuring less than 1/4 the distance between the xyphoid and the pubis, including laparoscopic surgery.
* Diagnosis of incisional hernia or presence of previous mesh on site.
* Midline laparotomy performed in less than 30 days.
* Pregnancy
* Severe trauma with hemodynamic instability
* Need for open abdomen or relaxing incisions
* Need for re-laparotomy during the first 30 postoperative days, except cases in which an abdominal wall dehiscence was diagnosed.
* Death during the first 30 postoperative days, except cases in which an abdominal wall dehiscence was diagnosed before the event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Fascial dehiscence incidence | 30 days

SECONDARY OUTCOMES:
Surgical site occurence (SSO) incidence | 30 days or during hospital stay
Surgical site occurrence requiring procedural intervention (SSOPI) incidence | 30 days or during hospital stay
Operative time (minutes), | 30 days
Hospital length of stay (days) | 30 days
Intensive care unit length of stay (days) | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez Diaz CJ, Rebasa Cladera P, Navarro Soto S, Hidalgo Rosas JM, Luna Aufroy A, Montmany Vioque S, Corredera Cantarin C. [Validation of abdominal wound dehiscence's risk model]. Cir Esp. 2014 Feb;92(2):114-9. doi: 10.1016/j.ciresp.2012.12.008. Epub 2013 May 3. Spanish. PMID 23648044
- [Result] van Ramshorst GH, Nieuwenhuizen J, Hop WC, Arends P, Boom J, Jeekel J, Lange JF. Abdominal wound dehiscence in adults: development and validation of a risk model. World J Surg. 2010 Jan;34(1):20-7. doi: 10.1007/s00268-009-0277-y. PMID 19898894
- [Derived] Lima HVG, Rasslan R, Novo FCF, Lima TMA, Damous SHB, Bernini CO, Montero EFS, Utiyama EM. Prevention of Fascial Dehiscence with Onlay Prophylactic Mesh in Emergency Laparotomy: A Randomized Clinical Trial. J Am Coll Surg. 2020 Jan;230(1):76-87. doi: 10.1016/j.jamcollsurg.2019.09.010. Epub 2019 Oct 28. PMID 31672681